CLINICAL TRIAL: NCT04087902
Title: A Prospective Longitudinal Quality of Life Study in Patients Undergoing Endoscopic Endonasal Skull Base Surgery
Brief Title: Long-Term Longitudinal QoL in Patients Undergoing EEA
Status: Recruiting | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Kyle Wu, Assistant Professor, Neurological Surgery, Ohio State University
Other Study IDs: 2019H0225
Record Dates: First submitted 2019-08-20; First posted 2019-09-12 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Pituitary Tumor; Meningioma; Rathke Cleft Cysts; Chordoma; Chondrosarcoma; Craniopharyngioma; Encephalocele; Esthesioneuroblastoma
Keywords: Endoscopic Endonasal Approach Surgery
MeSH Terms: conditions — Pituitary Neoplasms; Meningioma; Central Nervous System Cysts; Chordoma; Chondrosarcoma; Craniopharyngioma; Encephalocele; Esthesioneuroblastoma, Olfactory

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is a prospective longitudinal study to access postoperative 2-year quality of life in patients who undergo endonasal endoscopic approach surgeries of the skull base.

DETAILED DESCRIPTION:
This is a prospective single-institution longitudinal study to access quality of life in patients who undergo endonasal endoscopic approach surgeries of the skull base. Patients will be followed before surgery and up to twenty-four months post-surgery. The primary goal of the study is to assess the alterations to patient quality of life following endoscopic endonasal surgery using modern sinonasal reconstruction techniques. Secondary goals are to better understand the time course of normal healing and patient/procedural risk factors associated with poorer quality of life outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patient is scheduled to undergo endoscopic endonasal surgery. Multiple, staged surgeries are not exclusionary
* 18 years of age or older
* The subject must in the investigator's opinion, be psychosocially, mentally, and physically able to fully comply with this protocol including the required follow-up visits, the filling out of required forms, and have the ability to understand and give written informed consent

Exclusion Criteria:

* Patient is a prisoner
* Patient is not English speaking
* Patient is not expected to survive until the 2-year follow-up

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who are 18 years of age or older and undergoing surgery via Endoscopic Endonasal Approach.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-07-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
PROMIS-29 quality of life outcome measures for patients undergoing endoscopic endonasal surgeries. | 24-months post-operatively
  This study aims to better understand the long-term overall quality of life of patients undergoing endoscopic endonasal surgery using modern sinonasal reconstruction techniques. The PROMIS-29 metric, an overall quality of life metric, will be used to better understand quality of life for patients undergoing this procedure.

SECONDARY OUTCOMES:
ASK Nasal-12 questionnaire used to measure normal time of healing for patients undergoing endoscopic endonasal surgery | 24 months post-operatively
  This study aims to better understand the overall nose function in patients undergoing endoscopic endonasal surgery using modern sinonasal techniques. The ASK Nasal-12 metric is designed to evaluate nose overall nose function such as post-nasal drip, ability to smell, and pain.
Number of patients with long-term quality of life risk factors using PROMIS-29 | 24 months post-operatively
  This study aims to better understand the number of long-term risk factors for patients undergoing endoscopic endonasal surgeries using modern sinonasal reconstruction techniques. This will be done using the PROMIS-29 metric along with patient data.
Number of patients with long-term procedural comorbidities using ASK-Nasal 12. | 24 months post-operatively
  This study aims to better understand the number of long-term comorbidities for patients undergoing endonasal endoscopic surgeries using modern sinonasal reconstruction techniques. This will be done using the ASK-Nasal 12 metric along with patient data.

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Wu, MD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
There will be no sharing of individual participant data with other researchers. Data will be de-identified once analysis is complete and destroyed once manuscripts are written.